CLINICAL TRIAL: NCT04951869
Title: Assessing the Effectiveness of Protescal In Preventing Post Caesarean Section Hypertrophic Scar and Keloid
Brief Title: : Protescal: Prevention of Hypertrophic Scar and Keloid Formation Post Caesarean Section
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universiti Kebangsaan Malaysia Medical Centre (Other)
Responsible Party: Principal Investigator, Anizah Ali, Principle Investigator, Universiti Kebangsaan Malaysia Medical Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Research Code: FF-2017-170
Record Dates: First submitted 2021-05-30; First posted 2021-07-07 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-06

CONDITIONS: Caesarean Wound; Hypertrophic Surgical Scar; Keloid Scar Following Surgery
Keywords: caesarean section, hypertrophic scar, keloid, anti-adhesive gel, wound healing
MeSH Terms: conditions — Cicatrix, Hypertrophic; Keloid

STUDY DESIGN:
Intervention Model Description: concurrent 2 arms with study arm and control arm of women undergoing caesarean section without any previous abdominal surgeries
Who Masked: Participant
Masking Description: control group receives no protescal application while study group does
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Protescal group (Experimental): Caesarean-section was done in the usual manner. The transverse suprapubic skin incision was made and abdominal layers opened as usual. After delivering the baby, uterine muscle is closed in two layers with braided absorbable suture, polyglactin 910 (Vicryl no 1). After hemostasis secure, 1 mL Protescal gel was applied at the uterine suture site in Protescal group. Peritoneal layer closed using braided absorbable suture, polyglactin 910 (Vicryl no 1). Rectus sheath was sutured using braided absorbable suture, polyglactin 910 (Vicryl no 1). Subcutaneous tissue closed interruptedly using braided absorbable suture, polyglactin 910 (Vicryl no 1). Protescal gel (0.5 mL) was applied over the subcutaneous tissue prior to skin closure in Protescal group. The skin was then closed with the subcuticular method using braided absorbable suture, polyglactin 910 (Vicryl 3-0).
  Interventions: Drug: Protescal gel
- Control group (No Intervention): Caesarean-section was done in the usual manner. The transverse suprapubic skin incision was made and abdominal layers opened as usual. After delivering the baby, uterine muscle is closed in two layers with braided absorbable suture, polyglactin 910 (Vicryl no 1). After hemostasis secure, No Protescal gel was applied at the uterine suture site in this Control group. Peritoneal layer closed using braided absorbable suture, polyglactin 910 (Vicryl no 1). Rectus sheath was sutured using braided absorbable suture, polyglactin 910 (Vicryl no 1). Subcutaneous tissue closed interruptedly using braided absorbable suture, polyglactin 910 (Vicryl no 1). No application of Protescal gel (0.5 mL) over the subcutaneous tissue prior to skin closure in this Control group. The skin was then closed with the subcuticular method using braided absorbable suture, polyglactin 910 (Vicryl 3-0).

INTERVENTIONS:
Drug: Protescal gel — Protescal gel (0.5 mL) was again applied over the subcutaneous tissue prior to skin closure in Protescal group
  Arms: Protescal group

SUMMARY:
This study aimed to evaluate the effectiveness of Protescal in preventing post caesarean section hypertrophic scar and keloid formation.

DETAILED DESCRIPTION:
A randomized controlled trial was conducted for six months involving 90 women who underwent caesarean section without any history of previous abdominal surgery and who were planning for further pregnancy. They were randomized into two groups. The Protescal group was given Protescal gel which was applied over the uterine incision site and subcutaneous tissue layer prior to skin closure (n = 45), whereas in the control group, no Protescal gel was applied (n = 45). The primary outcome was to assess the healing of the external scar.

ELIGIBILITY:
Inclusion Criteria:

* All women undergoing elective caesarean section, without any history of previous abdominal surgery ; who planned for further pregnancy and consented to participate in this study.

Exclusion Criteria:

* Patient that allergic to protescal
* Patient with previous abdominal surgery
* Patient refusal or patients who are not able to give consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 90 (Actual)
Dates: Start 2017-04-26 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-11-16 (Actual)

PRIMARY OUTCOMES:
Name of the Measurement:Assessment of degree of caesarean wound healing. Measurement Tool:REEDA scale Unit of measure:"Percentage (%) of patients with..." | Day 10th post caesarean section
  Wound healing assessed on 10th-day post caesarean section using REEDA scale of which the criteria assessed include redness, edema, ecchymosis, discharge and approximation. The REEDA Scale (Redness, Edema, Ecchymosis, Discharge, Approximation) scale assesses the inflammation process and tissue healing. The minimum score is 0 and the maximum score is 15; whereby the higher the score denotes the more severe the tissue trauma and healing outcome.Percentage of patients in both groups with REEDA Scale scores of 0, 1-2 and ≥ 3 is determined.
Name of the Measurement : Assessment of Caesarean wound keloid formation & degree of scarring Measurement Tool : Modified Vancouver scar scale (MVSS) Unit of measure:"Percentage (%) of patients with..." | 3 months post caesarean section
  Third-month post-caesarean section, the degree of scarring was assessed using the Modified Vancouver scar scale (MVSS) which assessed pigmentation, height, pliability and vascularity of the scar. This scale focused on six parameters including scar height and thickness, pliability, vascularity, pigmentation, symptoms of itch and pain to generate a score ranging from 0 to 18 points.For the purpose of this study, a hypertrophic scar (HTS) was defined as one which was raised by at least 2 mm and had a total MVSS of 5 points or more (4). Thus a higher score would means a more hypertrophic scar formation. If a patient had more than one MVSS recorded during their follow up, the highest value was used.
Name of the Measurement : Assessment of Caesarean wound keloid formation & degree of scarring Measurement Tool : Colour photograph of wound Unit of measure : "Percentage (%) of patients with..." | 3 months post caesarean section
  Third-month post-caesarean section, the degree of scarring was assessed by colour photography if deemed necessary for comparison purposes. This would also depend on patient's agreement to her scar being photographed. If agreeable and deemed necessary, thus a patient's assessment was supplemented with colour photographs for later review and comparison.

SECONDARY OUTCOMES:
Name of the Measurement: Assessment of pelvic adhesions noted during next caesarean section.Measurement Tool: Intra-operative visual assesment of pelvic adhesions noted during next caesarean section.Unit of measure:"Percentage (%) of patients with..." | 3 years post caesarean section
  To assess the degree of pelvic adhesion formation intra-operatively during the next caesarean section. Visual assesment (by surgeons) of intra-operative findings of pelvic adhesions noted during next caesarean section which is documented in the intra-operative notes.

CONTACTS AND LOCATIONS:
Overall Officials: Anizah Ali, MD(UKM),MOG(UKM), Principal Investigator — UKMMC
Locations (1):
- Universiti Kebangsaan Malaysia Medical Centre, Cheras, Kuala Lumpur, Malaysia

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-04-26): https://cdn.clinicaltrials.gov/large-docs/69/NCT04951869/Prot_SAP_000.pdf
  • Informed Consent Form (2017-04-26): https://cdn.clinicaltrials.gov/large-docs/69/NCT04951869/ICF_001.pdf